CLINICAL TRIAL: NCT05247372
Title: The Effect of Iyengar Yoga Practice on Patients with Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Stanislav Machač, Ph.D, Principal Investigator, University Hospital, Motol
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK-809/21
Record Dates: First submitted 2022-01-03; First posted 2022-02-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Multiple Sclerosis, Iyenagar Yoga, Yoga, EDSS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The effect of Iyengar yoga practice on patients with multiple sclerosis (Other)
  Interventions: Other: The effect of Iyengar yoga practice on patients with multiple sclerosis

INTERVENTIONS:
Other: The effect of Iyengar yoga practice on patients with multiple sclerosis — The study will be conducted as a longitudinal follow-up - at first patients will fbe examined 2 months before the start of the exercise, than they will be examined at the beginning and end of the exercise, which they will attend for 3 months. Patients will be re-examined 2 months after the end of the exercise to clarify the continuing effect of the exercise. The examination will include a basic kinesiological analysis and a neurological examination,TUG test, 6MWT along with the Borg Subjective Weight Rating Scale and T25FWT, BBS, NHPT and stable sitting time in wheelchairs. To evaluate the development of the chest, the respiratory amplitude will be examined and the position of the spine in statics and dynamics will be evaluated using a spinal mouse. Quality of life will be assessed through the MFIS, MSIS-29, MSQOL 54 questionares and Beck's anxiety inventory.

SUMMARY:
The aim of this work is to find out what effect the practice of Iyengar yoga has on patients with multiple sclerosis on the EDSS 5 and more, specifically in the field of mobility, self-sufficiency and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* diagnosis of multiple sclerosis
* EDSS grade 5 or higher

Exclusion Criteria:

* age less than 18 years
* the patient is not diagnosed with multiple sclerosis EDSS grade less than 5
* refusal of the subject to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Hypothesis 1 | 3 months
  Increase in respiratory amplitud. It will be measured by the meter.
Hypothesis 2 | 3 months
  Increase in spinal development in the sagittal and frontal plane. It will by measured by spinal mouse.
Hypothesis 3 | 3 months
  Increase in walking speed measured by T25FWT. It will by measured by stopwatch.
Hypothesis 4 | 3 months
  Balance improvement in the Berg balance scale. It will be measured by the Berg balance scale questionare.
Hypothesis 5 | 3 months
  The quality of life of patients with MS is improved subjectively evaluated through MSQOL54 questionare.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Motol, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes